CLINICAL TRIAL: NCT04210401
Title: Registry of Culture Results From Reusable Duodenoscopes
Brief Title: Reusable Duodenoscope Culture Registry
Status: Withdrawn | Type: Observational
Why Stopped: Investigator did not move forward with the project due to costs.
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1513291
Record Dates: First submitted 2019-12-23; First posted 2019-12-24 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Duodenoscope Culture — Culture of reusable duodenoscopes following each use.

SUMMARY:
This project is being performed to examine the results of duodenoscope cultures following standard of care cleaning and reprocessing.

DETAILED DESCRIPTION:
This project is being performed to examine the results of duodenoscope cultures following standard of care cleaning and reprocessing. This information will allow us to elucidate the number of endoscopic procedures that can be performed using a single duodenoscope until microorganisms are cultured from duodenoscopes after standard of care cleaning and reprocessing. This will in turn allow us to improve the delivery of healthcare to patients undergoing endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Any patient undergoing endoscopic retrograde cholangiopancreatography procedure using a reusable duodenoscope

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data will be collected from patient who have a endoscopic retrograde cholangiopancreatography procedure at the Center for Interventional Endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Microorganism Growth | 6 months
  The aim of this registry is to identify the number of endoscopic procedures that can be performed using reusable duodenoscopes before microorganisms are grown from duodenoscope cultures following standard of care cleaning and reprocessing. This will enable us to identify the maximum number of procedures that can be performed with a single duodenoscope before being sent to the manufacturer to be refurbished.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth Orlando
Locations (1):
- Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No